CLINICAL TRIAL: NCT05413759
Title: Collaborative Pharmaceutical Care Initiated in Hospital and Continued in Primary Care to Improve Medication Adherence of Patients With Rheumatoid Arthritis
Brief Title: RhEumatoid Arthritis MEDIcation Adherence
Acronym: REMEDIA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 69HCL20_0272
Record Dates: First submitted 2022-05-23; First posted 2022-06-10 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Rheumatoid Arthritis
Keywords: medication adherence; rheumatoid arthritis; pharmaceutical care
MeSH Terms: conditions — Arthritis, Rheumatoid; Medication Adherence | interventions — Pharmaceutical Services

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pharmaceutical care in multiprofessional collaboration (Experimental): Medication reconciliation (hospital admission and discharge), disease-modifying antirheumatic drugs (DMARD) treatment information interview and 2 motivational interviews (after discharge, at 2 months and 6 months after the inclusion).
  Interventions: Other: Pharmaceutical care in multiprofessional collaboration
- Control group (usual practices group) (No Intervention): Usual follow-up during the 12-month follow-up.

INTERVENTIONS:
Other: Pharmaceutical care in multiprofessional collaboration — In addition to usual practices: medication reconciliation and pharmaceutical motivational interviews with patients (discharge, 2 & 6 months).
  Objective of medication reconciliation (admission): to detect and resolve unintended medication discrepancies between home medication list and treatment and hospital admission medication orders. Objective of medication reconciliation (discharge): to obtain an exact list of medication, to explain the medication modifications during hospitalization.
  Objective of the Disease-Modifying Antirheumatic Drugs information interview (discharge): to provide information and to answer questions on the management of treatment, to deal with practical situations to assess patients' self-management skills.
  Objective of interviews (2 & 6 months): to evaluate medications and their daily management, benefits and problems that patient may encounter, to assess the patient's ability to manage the treatment.
  Arms: Pharmaceutical care in multiprofessional collaboration

SUMMARY:
Rheumatoid arthritis (RA) is a public health issue because of its frequency, its functional consequences, the risk of morbidity and mortality and the costs incurred. A collaborative multiprofessional intervention initiated during hospitalization and continued after hospital discharge (ambulatory care ) would improve medication adherence in RA and therefore the health status of patients.

Main objective:

To compare, 12 months after the index hospitalization or consultation, the impact of pharmaceutical care provided in multiprofessional collaboration (pharmacist-physician) on medication adherence to disease-modifying treatments of patients with RA compared to usual care without pharmaceutical care and specific multi-professional collaboration.

Medication adherence to disease-modifying treatments will be assessed by the rate of coverage of disease-modifying treatments (or Medication Possession Ratio (MPR)).

METHODOLOGY: Interventional, multicenter, controlled, randomized, open label study, comparing in parallel 2 groups of patients with rheumatoid arthritis initially hospitalized in a rheumatology department (pharmaceutical care provided in multiprofessional collaboration (pharmacist-physician), initiated in the hospital and continued after hospital discharge (ambulatory care) vs traditional follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Patient with diagnosed rheumatoid arthritis (RA),
* Patient, male or female, aged 18 or over,
* Patient hospitalized or coming for a consultation in a rheumatology department, and returned home at hospital discharge
* Patient having DMARDs for RA (continuation or initiation) comprising at least methotrexate and/or a tsDMARD (targeted synthetic DMARD, JAK inhibitor) and/or subcutaneous bDMARD (biologic DMARD),
* Autonomous patient in the management of his drug treatment,
* Patient understanding and speaking French,
* Patient affiliated to the French general national health insurance or similar,
* Patient having given his free, informed and signed consent.

Exclusion Criteria:

* Patient whose usual pharmacy already has or has had a patient included in the INTERVENTION group in the study,
* Patient whose regular pharmacy is currently treating another patient.
* Patient with obvious significant cognitive or psychiatric disorders incompatible with the study (according to the judgment of the investigator),
* Patient whose management of his drug treatment at home is carried out exclusively by a carer,
* Patient participating in another research that may interfere (investigator's judgement) with the results of the present study,
* Adult patient protected under the terms of the law (Public Health Code),
* Patient not fit to carry out the follow-up, according to the judgment of the investigator,
* Pregnant or breastfeeding women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2022-06-28 (Actual); Primary Completion 2026-12-28 (Estimated); Study Completion 2027-12-28 (Estimated)

PRIMARY OUTCOMES:
Medication adherence to rheumatoid arthritis treatment | Month 12
  The primary endpoint is the rate of adherent patients to DMARDs after 12 months of follow-up assessed by the Medication Possession Ratio (MPR).
  The MPR is calculated for each drug: total quantity of dose units dispensed compared to the theoretical quantity of dose units necessary for compliance with the prescribed dosage. The calculation will be made from:
  * dispensing data collected from the patient's community pharmacist (control and intervention group),
  * prescription data from all prescriptions (between Month 0 and Month 12), reported by the patient during the visit to Month 12,
  * and hospitalization data from the medicalized information system program (PMSI:) and the patient log.
  A patient is considered adherent to his treatment if the MPR is greater than or equal to 80%. For patients with more than one DMARD drug prescribed, they will be considered adherent if the MPR of each DMARD is greater than or equal to 80%.

SECONDARY OUTCOMES:
Clinical criteria - Evolution of the Disease Activity Score DAS28 | Day 0 and Month 12
  A Disease Activity Score (DAS) indicates the severity of rheumatoid arthritis disease activity at a given moment in time. It is calculated based on several different factors, including lab results, patient feedback, and joint swelling and tenderness.
  A traditional DAS score requires examining 44 specific joints.
  The DAS28 score is arrived at using:
  The number of swollen joints (out of the 28), The number of tender joints (out of the 28), The C reactive protein (CRP) or erythrocyte sedimentation rate (ESR) lab test results Answers to a patient health assessment questionnaire A mathematical formula is used to calculate the overall score. DAS28 can range from 0 to 9.4.
  Generally, a DAS28 score of:
  More than 5.1 indicates high disease activity Between 3.2 and 5.1 indicates moderate disease activity Between 2.6 and less than 3.2 indicates low disease activity Lower than 2.6 indicates disease remission
Clinical criteria - Number of Rheumatoid Arthritis-related re-hospitalizations | Month 0 and Month 12
  Number of Rheumatoid Arthritis-related re-hospitalizations between Month 0 and Month 12
Clinical criteria - Number of adverse effects related to drug treatments leading to hospitalization. | Month 0 and Month 12
  Number of adverse effects related to drug treatments leading to hospitalization between Month 0 and Month 12.
Functional and quality of life criteria - Evolution of the Health Assessment Questionnaire (HAQ) score | Day 0 and Month 12
  The Evolution of the Health Assessment Questionnaire (HAQ) is an 24-item questionnaire.
  Each question is assigned the following score:
  0 = without any difficulty ; 1 = with some difficulty ; 2 = with great difficulty ; 3 = unable to do so The rating for each of the 8 domains is the one corresponding to the highest score for the questions in that domain.
  The notion of need for help from a third person and/or use of devices can modify this rating system. In this case, the score for the area concerned must be at least equal to 2.
  The functional index is the sum of the ratings of the various domains divided by the number of domains evaluated (normally 8, but less in case of totally missing data for a particular domain).
  The score obtained is between 0 and 3. The higher the score, the more disabling the pathology.
Functional and quality of life criteria - Evolution of the EuroQol 5-Dimensional score (EQ-5D) | Day 0 and Month 12
  The EuroQol 5-Dimensional score (EQ-5D) is a standardised measure of health-related quality of life.
  The EQ-5D descriptive system comprises five dimensions: mobility, self-care, usual activities, pain and discomfort, and anxiety and depression.
  The evaluation component requires a patient to record their overall health status using a visual analogue scale (EQ-VAS).
  Following assessment the scores from the descriptive component can be reported as a five digit number ranging from 11111 (full health) to 33333/55555 (worst health). A number of methods exist for analysing these five digit profiles. Frequently they are converted to a single utility index using country specific value sets, which can be used in the clinical and economic evaluation of health care as well as in population health surveys.
Criteria for patient behavior in relation to their disease-modifying antirheumatic drugs (DMARDs) - Medication Possession Ratio for each disease-modifying antirheumatic drug (DMARD) | Month 12
  The Medication Possession Ratio is calculated for each drug: total quantity of dose units dispensed compared to the theoretical quantity of dose units necessary for compliance with the prescribed dosage. The calculation will be made from:
  * dispensing data collected from the patient's community pharmacist (control and intervention group),
  * prescription data from all prescriptions (between Month 0 and Month 12), reported by the patient during the visit to Month 12,
  * and hospitalization data from the medicalized information system program (PMSI:) and the patient log.
Criteria for patient behavior in relation to their disease-modifying antirheumatic drugs (DMARDs) - Adherent rate according to the Compliance Questionnaire on Rheumatology (CQR) | Month 12
  The Compliance Questionnaire on Rheumatology (CQR) is a 19 item, self-administered questionnaire that was developed with the aim of correctly identifying patients that were classified as "low" adhering participants (taking <80% of their medication correctly). The four point Likert answering scale ranges from; "Definitely don't agree" (scored 1) to "Definitely agree" (scored 4) with lower scores indicating lower levels of adherence.
Criteria for patient behavior in relation to their disease-modifying antirheumatic drugs (DMARDs) - Evolution of the BioSecure score or Knowledge score (Methotrexate and/or anti-JAK) | Day 0 and Month 12
  The BioSecure questionnaire assess self-management skills and knowledge and patient safety under biotherapy. It has 55 questions regarding 24 areas of competence. The final score is between 0 and 100, a high score reflecting better knowledge.
  Questionnaire about Methotrexate assess self-management skills and knowledge and patient safety under Methotrexate. It has 7 questions and 1 scenario (to be chosen by the doctor out of 5). One point is awarded for each correct answer (refer to the correction of the questionnaire). Total out of 100: (score x 100)/ 31. The final score is between 0 and 100, a high score reflecting better knowledge.
  Questionnaire about anti-JAK assess self-management skills and knowledge and patient safety under anti-JAK. It has 8 questions and 6 scenario. One point is awarded for each correct answer (refer to the correction of the questionnaire). Total out of 100: sum x 1.92. The final score is between 0 and 100, a high score reflecting better knowledge.
Criteria for patient behavior in relation to their disease-modifying antirheumatic drugs (DMARDs) - Evolution of the Beliefs about Medicines Questionnaire (BMQ) score | Day 0 and Month 12
  The BMQ consists of two five-item scales assessing patients' beliefs about the necessity of prescribed medication for controlling their disease and their concerns about potential adverse consequences of taking it. Respondents indicate their degree of agreement with each statement on a five-point Likert scale, ranging from 1 = strongly disagree to 5 = strongly agree. Scores obtained for individual items within both scales are summed. Thus, total scores for the Necessity and Concerns Scales range from 5 to 25. Higher scores indicate stronger beliefs.
Economic criterion | Month 12
  Costs of managing the two strategies.
Intervention implementation and acceptability criteria - Satisfaction of pharmacists and general practitioners through semi-structured interviews | Month 12
  Satisfaction of pharmacists and general practitioners through semi-structured interviews at Month 12
Intervention implementation and acceptability criteria - Duration of follow-up interviews measured by community pharmacist | Month 2 and Month 6
  Duration of follow-up interviews measured by community pharmacist at Month 2 and Month 6
Intervention implementation and acceptability criteria - Number of patients having benefited from a complete follow-up by the town pharmacist (participation in the 2 scheduled meetings to reinforce medication adherence) | Month 12
  Number of patients having benefited from a complete follow-up by the town pharmacist (participation in the 2 scheduled meetings to reinforce medication adherence)
Intervention implementation and acceptability criteria - Patient satisfaction by questionnaire | Month 12
  Patient satisfaction assessed by a 6_item questionnaire completed by patients in the interventional group.
  The 6 items are rated on a 4-dimension Likert-scale : "Not at all satisfied", "Not very satisfied", "Quite satisfied", "Completely satisfied". Answers will be the subject of a descriptive analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Roland CHAPURLAT, MD/PHD, Principal Investigator — Hospices Civils de Lyon
Locations (2):
- France (2):
  - Service de rhumatologie, Centre Hospitalier Lyon Sud, Groupement Hospitalier Sud, Hospices Civils de Lyon, Pierre-Bénite, Lyon
  - Service de rhumatologie et pathologie osseuse - Hôpital Edouard Herriot, Lyon

IPD SHARING:
Plan to Share IPD: No